CLINICAL TRIAL: NCT00740948
Title: Tolerance and Efficacy of Rituximab in Sjogren's Disease
Acronym: TEARS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TEARS
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Sjogren's Disease
Keywords: Sjogren's disease; Rituximab; Treatment; anti CD20
MeSH Terms: conditions — Sjogren's Syndrome | interventions — Rituximab; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Rituximab
  Interventions: Drug: Rituximab (mabthera) Injection
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo: NaCl 0.9% or Glucose 5%

INTERVENTIONS:
Drug: Rituximab (mabthera) Injection — 2 * 1g of Rituximab at the 1st day and at the 14th day.
  Arms: 1
Drug: Placebo: NaCl 0.9% or Glucose 5% — 2* 250ml of NaCl 0.9% or Glucose 5% at the 1st day and at the 14th day.
  Arms: 2

SUMMARY:
CLINICAL PHASE II INDICATION Sjogren's syndrome RATIONALE Sjögren's syndrome (SS) is an autoimmune disorder affecting 0.2% to 3% of the general population. Pharmacological treatment can improve the sicca symptoms, often transiently, but they are unable to modify the course of the disease.Open label studies suggested that low-dose rituximab produced acute and complete CD20 depletion in blood and tissue; was well tolerated without corticosteroid use; and significantly improved glandular and extra-glandular manifestations of pSS. Larger controlled studies are now warranted. Our hypothesis is that two infusions of 1000 mg of Rituximab may be better than placebo to treat patients suffering from pSS. To test this hypothesis, we propose to compare patients with recent and/or severe pSS treated with either Rituximab or placebo.

OBJECTIVES Primary objective : Evaluation of the efficacy defined as a 30% improvement between Day 1 and Week 24 in the values on 2 of the 4 VAS measuring global scores of the disease (activity of the disease including extra glandular manifestations), joint pain, fatigue, and the most disturbing dryness.Secondary objectives : Variations from baseline to week 24 of:

The 0-100-mm VAS scores for dry mouth, dry eyes, dry trachea, dry vagina, and dry skin; fatigue; pain; Tender and swollen joint counts; Tender points; Other systemic manifestation; Unstimulated salivary flow rate; Schirmer and van Bijsterveld scores (2-3); C-reactive protein (CRP) and erythrocyte sedimentation rate (ESR); rheumatoid factor (RF); ANA; serum IgG, IgA, and IgM; complement; cryoglobulinemia; and counts of B and T cells; Evaluation of the safety of Rituximab during the study Evaluation of the improvement evaluated on VAS by the physician Evaluation of the disease activity scores as suggested by Bowman and Vitali Evaluation of Chisholm score, B cells characteristics and DNA microarray on labial accessory salivary gland (SG) biopsy samples, and salivary gland echography at inclusion and at week 24.

TRIAL DESIGN Multicenter, randomized, double-blind, placebo-controlled trial NUMBER OF SUBJECTS : 120

DETAILED DESCRIPTION:
TARGET POPULATION Inclusion criteria : Patients will be eligible if :

they fulfill the new American-European Consensus Group criteria for pSS and have :

* a recent (less than 10 years) and active disease as assessed by :
* values > 50 mm on 2 of 4 visual analogue scales (VAS) (0-100mm) that evaluated global scores of the disease (activity of the disease including extra glandular manifestations), pain, sicca syndrome and fatigue over the last week.
* Rheumatoid factor or SSA>1.5N or cryoglobulinemia or hypergammaglobulinemia or high level of beta2 microglobulinemia or hypocomplémentemia.
* and/or at least one of the following severe signs: parotidomegaly, arthritis, purpura, pulmonary involvement, tubulopathy, neurological involvement, thrombocytopenia.

Additional inclusion criteria will be as follows:

* informed consent
* age 18-80 years,
* stable non-steroidal anti-inflammatory drugs
* and no prescription of immunosuppressive agents for at least 4 weeks prior to inclusion
* Use of a reliable mean of contraception (for patients of reproductive potential)

Exclusion criteria :

Patients should be excluded if they have a secondary SS, if they received cytotoxic drugs during the previous 4 months, if they have severe renal or haematological failure, a history of cancer, hepatitis B or C, HIV, tuberculosis, severe diabetes or any other chronic disease or evidence of infection, if they have had severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies or if they are unable to understand the protocol. Other : neutrophil count < 1.5 x 103/L, live/attenuated vaccine within 28 days prior to baseline, pregnancy, breast feeding,

ELIGIBILITY:
Inclusion Criteria:

* they fulfill the new American-European Consensus Group criteria for pSS and have :
* a recent (less than 10 years) and active disease as assessed by :
* values > 50 mm on 2 of 4 visual analogue scales (VAS) (0-100mm) that evaluated global scores of the disease (activity of the disease including extra glandular manifestations), pain, sicca syndrome and fatigue over the last week.
* Rheumatoid factor or anti SSA>1.5N or cryoglobulinemia or
* hypergammaglobulinemia or high level of beta2 microglobulinemia or
* hypocomplémentemia.
* and/or at least one of the following severe signs:

  * parotidomegaly,
  * arthritis,
  * purpura,
  * pulmonary involvement,
  * tubulopathy,
  * neurological involvement,

informed consent age 18-80 years, stable non-steroidal anti-inflammatory drugs and no prescription of immunosuppressive agents for at least 4 weeks prior to inclusion Use of a reliable mean of contraception (for patients of reproductive potential)

Exclusion Criteria:

* Patients should be excluded if they have a secondary SS,
* if they received cytotoxic drugs during the previous 4 months,
* if they have severe renal or haematological failure, a history of cancer, hepatitis B or C, HIV, tuberculosis, severe diabetes or any other chronic disease or evidence of infection,
* if they have had severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* or if they are unable to understand the protocol.
* Other : neutrophil count < 1.5 x 103/L, live/attenuated vaccine within 28 days prior to baseline, pregnancy, breast feeding,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2008-03; Primary Completion 2012-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
30% improvement between in the values on 2 of the 4 VAS measuring global scores of the disease (activity of the disease), joint pain, fatigue, and dryness. | 24 weeks

SECONDARY OUTCOMES:
Variations from baseline to week 24 of clinical, biological and histological data | 24, 36 and 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alain SARAUX, Pr, Principal Investigator — University Hospital, Brest
Locations (14):
- France (14):
  - CHU de Brest, Brest
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - GH Le Havre, Le Havre
  - AP-HP Bicêtre, Le Kremlin-Bicêtre
  - Ch Le Mans, Le Mans
  - CHRU de LILLE, Lille
  - CHU de Marseille, Marseille
  - Hopital LAPEYRONIE, Montpellier
  - CHU de Nantes, Nantes
  - Hôpital Cochin APHP, Paris
  - CHU Bichat, Paris
  - Hôpital SUD CHU Rennes, Rennes
  - CHU Rouen, Rouen
  - CHU de Strasbourg, Strasbourg

REFERENCES:
- [Background] Devauchelle-Pensec V, Pennec Y, Morvan J, Pers JO, Daridon C, Jousse-Joulin S, Roudaut A, Jamin C, Renaudineau Y, Roue IQ, Cochener B, Youinou P, Saraux A. Improvement of Sjogren's syndrome after two infusions of rituximab (anti-CD20). Arthritis Rheum. 2007 Mar 15;57(2):310-7. doi: 10.1002/art.22536. PMID 17330280
- [Derived] Cornec D, Devauchelle-Pensec V, Mariette X, Jousse-Joulin S, Berthelot JM, Perdriger A, Puechal X, Le Guern V, Sibilia J, Gottenberg JE, Chiche L, Hachulla E, Yves Hatron P, Goeb V, Hayem G, Morel J, Zarnitsky C, Dubost JJ, Saliou P, Pers JO, Seror R, Saraux A. Severe Health-Related Quality of Life Impairment in Active Primary Sjogren's Syndrome and Patient-Reported Outcomes: Data From a Large Therapeutic Trial. Arthritis Care Res (Hoboken). 2017 Apr;69(4):528-535. doi: 10.1002/acr.22974. PMID 27390310
- [Derived] Costa S, Schutz S, Cornec D, Uguen A, Quintin-Roue I, Lesourd A, Berthelot JM, Hachulla E, Hatron PY, Goeb V, Vittecoq O, Pers JO, Marcorelles P, Saraux A, Devauchelle-Pensec V. B-cell and T-cell quantification in minor salivary glands in primary Sjogren's syndrome: development and validation of a pixel-based digital procedure. Arthritis Res Ther. 2016 Jan 20;18:21. doi: 10.1186/s13075-016-0924-2. PMID 26785742
- [Derived] Jousse-Joulin S, Devauchelle-Pensec V, Cornec D, Marhadour T, Bressollette L, Gestin S, Pers JO, Nowak E, Saraux A. Brief Report: Ultrasonographic Assessment of Salivary Gland Response to Rituximab in Primary Sjogren's Syndrome. Arthritis Rheumatol. 2015 Jun;67(6):1623-8. doi: 10.1002/art.39088. PMID 25708147
- [Derived] Devauchelle-Pensec V, Mariette X, Jousse-Joulin S, Berthelot JM, Perdriger A, Puechal X, Le Guern V, Sibilia J, Gottenberg JE, Chiche L, Hachulla E, Hatron PY, Goeb V, Hayem G, Morel J, Zarnitsky C, Dubost JJ, Pers JO, Nowak E, Saraux A. Treatment of primary Sjogren syndrome with rituximab: a randomized trial. Ann Intern Med. 2014 Feb 18;160(4):233-42. doi: 10.7326/M13-1085. PMID 24727841